CLINICAL TRIAL: NCT06961006
Title: A Phase 2, Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled Clinical Study of V940 (mRNA-4157) Plus Pembrolizumab Versus Placebo Plus Pembrolizumab in Participants With First-Line Advanced Melanoma (INTerpath-012)
Brief Title: A Clinical Study of V940 and Pembrolizumab (MK-3475) in People With Melanoma (V940-012/INTerpath-012)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V940-012; V940-012 (Other: MSD); INTerpath-012 (Other: MSD); 2023-504923-20-00 (Registry Identifier: EU CT); U1111-1290-3969 (Registry Identifier: UTN)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Malignant Melanoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V940 + Pembrolizumab (Experimental): Participants will receive 1 mg of V940 via intramuscular (IM) injection every 3 weeks (q3w) for up to 9 doses (up to approximately 27 weeks) plus 400 mg of pembrolizumab via intravenous (IV) infusion every 6 weeks (q6w) for up to 17 doses, or for a total treatment duration of up to approximately 2 years, or until disease progression or discontinuation.
  Interventions: Biological: V940; Biological: Pembrolizumab
- Placebo + Pembrolizumab (Active Comparator): Participants will receive placebo via IM injection q3w for up to 9 doses (up to approximately 27 weeks) plus 400 mg of pembrolizumab via IV infusion q6w for up to 17 doses, or for a total treatment duration of up to approximately 2 years, or until disease progression or discontinuation.
  Interventions: Biological: Pembrolizumab; Other: Placebo

INTERVENTIONS:
Biological: V940 — IM injection
  Other Names: mRNA-4157
  Arms: V940 + Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Other: Placebo — IM injection
  Arms: Placebo + Pembrolizumab

SUMMARY:
Researchers want to learn if V940 with pembrolizumab can stop advanced melanoma from growing or spreading. Melanoma is a type of skin cancer. Advanced means the cancer has spread to other parts of the body and cannot be removed with surgery. A standard (or usual) treatment for advanced melanoma is immunotherapy. Immunotherapy is a treatment that helps the immune system fight cancer. V940 is a study treatment designed to help a person's immune system attack their specific cancer. Pembrolizumab is an immunotherapy.

The goal of this study is to learn if people who receive V940 with pembrolizumab live longer without the cancer growing or spreading than people who receive placebo with pembrolizumab. A placebo looks like the study treatment but has no study treatment in it. Using a placebo helps researchers better understand the effects of a study treatment.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has unresectable and histologically confirmed Stage III or IV cutaneous melanoma per American Joint Committee on Cancer (AJCC) Eighth Edition guidelines.
* Has been untreated for melanoma except if participant received prior adjuvant or neoadjuvant therapy with targeted therapy or immunotherapy (such as anti-cytotoxic T-lymphocyte-associated protein [CTLA-4], anti-programmed cell death 1 protein [PD-1] therapy or interferon), and only if relapse did not occur within 12 months after treatment discontinuation.
* Have documentation of serine/threonine-protein kinase B-raf (BRAF) V600-activating mutation status or had BRAF V600 mutation testing per local institutional standards during the screening period (participants with BRAF mutation positive melanoma as well as BRAF wild-type or unknown are eligible).
* Have the presence of at least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as determined by the local site investigator/radiology assessment.
* Provides tumor tissue (preferably from a metastatic site and, if not available, from the primary tumor) that is suitable for next generation sequencing and biomarker analysis as required for this study.
* Participants with human immunodeficiency virus (HIV) must have well controlled HIV on antiretroviral therapy (ART).
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has clinically significant heart failure, defined as New York Heart Association class III or IV, within the past 6 months, unless the disease is well controlled in the opinion of the investigator.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has ocular or mucosal melanoma.
* Received transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 2 weeks of the Screening blood sample (including the blood sample for V940 generation).
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, lymphocyte activation gene 3 [LAG-3], tumor necrosis factor receptors [OX-40 or CD137]), with some exceptions.
* Received prior systemic anticancer therapy for melanoma before randomization, with some exceptions.
* Received prior radiotherapy within 2 weeks of start of study intervention or has ongoing radiation related toxicities.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Received prior treatment with another universal or personalized cancer vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2028-07-22 (Estimated); Study Completion 2031-09-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by investigator assessment or death due to any cause, whichever occurs first. Progressive disease (PD) is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS per RECIST 1.1 as assessed by investigator will be presented.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 6 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR per RECIST 1.1 as assessed by investigator will be presented.
Duration of Response (DOR) | Up to approximately 6 years
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by investigator will be presented.
Overall Survival (OS) | Up to approximately 6 years
  OS is defined as time from randomization to death due to any cause.
Number of Participants With ≥1 Adverse Event (AE) | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience one or more AEs will be reported.
Number of Participants Discontinuing From Study Therapy Due to AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (37):
- United States (5):
  - Highlands Oncology Group ( Site 4042), Springdale, Arkansas
  - UCSF Medical Center at Mission Bay ( Site 4044), San Francisco, California
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 4047), Hackensack, New Jersey
  - Inova Schar Cancer Institute ( Site 4046), Fairfax, Virginia
  - Fred Hutchinson Cancer Center ( Site 4041), Seattle, Washington
- Australia (3):
  - Blacktown Hospital ( Site 2001), Blacktown, New South Wales
  - Melanoma Institute Australia ( Site 2000), Wollstonecraft, New South Wales
  - One Clinical Research ( Site 2002), Nedlands, Western Australia
- William Osler Health System (Brampton Civic Hospital) ( Site 2023), Brampton, Ontario, Canada
- France (3):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Dermatology Department ( Site 2042), Nice, Alpes-Maritimes
  - Hôpital Saint-Louis ( Site 2041), Paris, Île-de-France Region
  - Gustave Roussy ( Site 2040), Villejuif, Île-de-France Region
- Germany (5):
  - NCT ( Site 2065), Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt Goethe-Universität ( Site 2063), Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln ( Site 2064), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 2061), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 2060), Hamburg
- Greece (3):
  - General Hospital of Athens "Laiko" ( Site 2080), Athens, Attica
  - Metropolitan Hospital ( Site 2082), Athens, Attica
  - European Interbalkan Medical Center ( Site 2081), Thessaloniki
- Israel (4):
  - Emek Medical Center ( Site 3003), Afula
  - Hadassah Medical Center ( Site 3001), Jerusalem
  - Rabin Medical Center ( Site 3002), Petah Tikva
  - Sheba Medical Center ( Site 3000), Ramat Gan
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 3021), Milan, Milano
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 3020), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 3022), Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 3023), Roma
- Harbour Cancer & Wellness ( Site 3040), Auckland, New Zealand
- Poland (2):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 3061), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 3060), Warsaw, Masovian Voivodeship
- Portugal (3):
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 4002), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 4001), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 4000), Porto
- Spain (3):
  - Hospital Universitari Vall d'Hebron ( Site 3081), Barcelona
  - Hospital Clínic Barcelona ( Site 3080), Barcelona
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 3082), Madrid

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/